CLINICAL TRIAL: NCT00436007
Title: Safety and Immunogenicity Study of GSK Biologicals' Investigational Vaccination Regimen Malaria Vaccine 257049, When Incorporated Into an Expanded Program on Immunization (EPI) Regimen That Includes Tritanrix HepB/Hib, OPV, Measles and Yellow Fever Vaccination in Infants
Brief Title: Safety and Immunogenicity Study of GSK Biologicals' Malaria Vaccine 257049, When Incorporated Into an EPI Regimen
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 106369
Record Dates: First submitted 2007-02-15; First posted 2007-02-16 (Estimated); Results first posted 2013-05-27 (Estimated); Last update posted 2018-08-16 (Actual); Status verified 2017-04

CONDITIONS: Malaria
Keywords: Africa; Plasmodium falciparum; Malaria
MeSH Terms: conditions — Malaria; Malaria, Falciparum | interventions — RTS malaria vaccine; Yellow Fever Vaccine; Poliovirus Vaccine, Oral

ARMS (3):
- GSK 257049 1 Group (Experimental): Subjects aged 6 to 10 weeks at the time of first vaccination received 3 doses of Tritanrix™ HepB/Hib, Polio Sabin™ and GSK 257049 vaccines at Months 0, 1 and 2, and a single dose of Rouvax™ and Stamaril™ vaccines at Month 7.
  The GSK 257049 and Tritanrix™ HepB/Hib vaccines were administered intramuscularly in the left and right antero-lateral thigh, respectively. Rouvax™ and Stamaril™ were administered intramuscularly in the left and right arm respectively. Polio Sabin™ was administered orally. The Stamaril™ vaccine was not administered to subjects from Tanzania as this vaccine was not foreseen at the time to be introduced to the EPI vaccination schedule in Tanzania.
  Interventions: Biological: GSK 257049; Biological: Tritanrix™ HepB/Hib; Biological: Rouvax™; Biological: Stamaril™; Biological: Polio Sabin™
- GSK 257049 2 Group (Experimental): Subjects aged 6 to 10 weeks at the time of first vaccination received 3 doses of Tritanrix™ HepB/Hib and Polio Sabin™ at Months 0, 1 and 2, 3 doses of GSK 257049 vaccine at Months 0, 1 and 7, and a single dose of Rouvax™ and Stamaril™ at Month 7. The GSK 257049 and Tritanrix™ HepB/Hib vaccines were administered intramuscularly in the left and right antero-lateral thigh, respectively. Rouvax™ and Stamaril™ were administered intramuscularly in the left and right arm respectively. Polio Sabin™ was administered orally. Stamaril™ was not administered to subjects from Tanzania as this vaccine was not foreseen at the time to be introduced to the EPI vaccination schedule in Tanzania.
  Interventions: Biological: GSK 257049; Biological: Tritanrix™ HepB/Hib; Biological: Rouvax™; Biological: Stamaril™; Biological: Polio Sabin™
- Tritanrix™ HepB/Hiberix™ Group (Active Comparator): Subjects aged 6 to 10 weeks at the time of first vaccination received 3 doses of Tritanrix™ HepB/Hib and Polio Sabin™ at Months 0, 1 and 2, and a single dose of Rouvax™ and Stamaril™ at Month 7. The GSK 257049 and Tritanrix™ HepB/Hib vaccines were administered intramuscularly in the left and right antero-lateral thigh, respectively. Rouvax™ and Stamaril™ were administered intramuscularly in the left and right arm respectively. Polio Sabin™ was administered orally. The Stamaril™ vaccine was not administered to subjects from Tanzania as this vaccine was not foreseen at the time to be introduced to the EPI vaccination schedule in Tanzania.
  Interventions: Biological: Tritanrix™ HepB/Hib; Biological: Rouvax™; Biological: Stamaril™; Biological: Polio Sabin™

INTERVENTIONS:
Biological: GSK 257049 — GlaxoSmithKline (GSK) Biologicals' candidate Plasmodium falciparum malaria vaccine
  Arms: GSK 257049 1 Group; GSK 257049 2 Group
Biological: Tritanrix™ HepB/Hib — GSK Biologicals' re-constituted diphtheria, tetanus, pertussis, hepatitis B vaccine (Tritanrix™ HepB) and Haemophilus influenzae type B vaccine (Hiberix™)
  Other Names: DTPwHepB/Hib vaccine
Biological: Rouvax™ — Aventis Pasteur's attenuated measles vaccine.
Biological: Stamaril™ — Aventis Pasteur's attenuated yellow fever vaccine.
  Other Names: Yellow Fever Vaccine
Biological: Polio Sabin™ — GSK Biologicals' oral polio virus vaccine
  Other Names: Oral Polio vaccine (OPV).

SUMMARY:
This study is being done to assess the possibility of the potential integration of malaria vaccine into the EPI regimen. It will evaluate whether the malaria vaccine is safe and immunogenic in infants aged 6 to 10 weeks at first dose, when co-administered with other EPI vaccine antigens. The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

DETAILED DESCRIPTION:
Two vaccination schedules will be studied, which constitutes the two alternative three dose regimens for the malaria candidate vaccine 257049 integration into EPI. The co-administered EPI vaccines include GSK Biologicals' Tritanrix™-HepB/Hiberix™, a measles vaccine (depending on the supply availability), Aventis Pasteur's Yellow Fever vaccine Stamaril™ and GSK Biologicals' Oral Polio vaccine Polio Sabin™. Tuberculosis vaccine (Bacillus of Calmette and Guerin, BCG) will be administered according to national medical practice and will not be administered as part of this protocol, but will be documented.

ELIGIBILITY:
Inclusion Criteria:

* A male or female infant between 6 and 10 weeks of age at the time of first vaccination.
* Signed or thumb-printed informed consent obtained from the parent(s)/guardian(s) of the child. Where parent(s)/guardian(s) are illiterate, the consent form will be countersigned by a witness.
* Subjects who have received one previous dose of OPV and BCG.
* Subjects who are born after a normal gestation period (between 36 and 42 weeks).

Exclusion Criteria:

* Acute disease at the time of enrolment.
* Serious acute or chronic illness determined by clinical or physical examination and laboratory screening tests.
* Laboratory screening tests out of range, specifically: ALT and creatinine above acceptable limit; Hemoglobin, Platelet count and Total white cell count below acceptable limit.
* Previous vaccination with diphtheria, tetanus, pertussis (whole-cell or acellular), Hemophilus influenzae type b or hepatitis B vaccines.
* BCG administration within one week of proposed administration of a study vaccine.
* OPV administration within four weeks of proposed administration of a study vaccine.
* Planned administration/administration of a vaccine not foreseen by the study protocol within 30 days of the first dose of vaccine(s).
* Use of any investigational or non-registered drug or vaccine within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Administration of immunoglobulins, blood transfusions or other blood products since birth to the first dose of study vaccine or planned administration during the study period.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Simultaneous participation in any other clinical trial.
* Twins (to avoid misidentification).
* Maternal death.
* History of allergic reactions (significant IgE-mediated events) or anaphylaxis to previous immunizations.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Any other findings that the investigator feels would increase the risk of having an adverse outcome from participation in the trial.

Ages: 6 Weeks to 10 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 511 (Actual)
Dates: Start 2007-04-30; Primary Completion 2008-09-15 (Actual); Study Completion 2009-10-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- GSK Investigational Site, Lambaréné, Gabon
- GSK Investigational Site, Kintampo, Ghana
- GSK Investigational Site, Dar es Salaam, Tanzania

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Ajua A, Lell B, Agnandji ST, Asante KP, Owusu-Agyei S, Mwangoka G, Mpina M, Salim N, Tanner M, Abdulla S, Vekemans J, Jongert E, Lievens M, Cambron P, Ockenhouse CF, Kremsner PG, Mordmuller B. The effect of immunization schedule with the malaria vaccine candidate RTS,S/AS01E on protective efficacy and anti-circumsporozoite protein antibody avidity in African infants. Malar J. 2015 Feb 13;14:72. doi: 10.1186/s12936-015-0605-7. PMID 25885325
- [Derived] Warimwe GM, Fletcher HA, Olotu A, Agnandji ST, Hill AV, Marsh K, Bejon P. Peripheral blood monocyte-to-lymphocyte ratio at study enrollment predicts efficacy of the RTS,S malaria vaccine: analysis of pooled phase II clinical trial data. BMC Med. 2013 Aug 21;11:184. doi: 10.1186/1741-7015-11-184. PMID 23962071
- [Derived] Asante KP, Abdulla S, Agnandji S, Lyimo J, Vekemans J, Soulanoudjingar S, Owusu R, Shomari M, Leach A, Jongert E, Salim N, Fernandes JF, Dosoo D, Chikawe M, Issifou S, Osei-Kwakye K, Lievens M, Paricek M, Moller T, Apanga S, Mwangoka G, Dubois MC, Madi T, Kwara E, Minja R, Hounkpatin AB, Boahen O, Kayan K, Adjei G, Chandramohan D, Carter T, Vansadia P, Sillman M, Savarese B, Loucq C, Lapierre D, Greenwood B, Cohen J, Kremsner P, Owusu-Agyei S, Tanner M, Lell B. Safety and efficacy of the RTS,S/AS01E candidate malaria vaccine given with expanded-programme-on-immunisation vaccines: 19 month follow-up of a randomised, open-label, phase 2 trial. Lancet Infect Dis. 2011 Oct;11(10):741-9. doi: 10.1016/S1473-3099(11)70100-1. Epub 2011 Jul 22. PMID 21782519
- [Derived] Agnandji ST, Asante KP, Lyimo J, Vekemans J, Soulanoudjingar SS, Owusu R, Shomari M, Leach A, Fernandes J, Dosoo D, Chikawe M, Issifou S, Osei-Kwakye K, Lievens M, Paricek M, Apanga S, Mwangoka G, Okissi B, Kwara E, Minja R, Lange J, Boahen O, Kayan K, Adjei G, Chandramohan D, Jongert E, Demoitie MA, Dubois MC, Carter T, Vansadia P, Villafana T, Sillman M, Savarese B, Lapierre D, Ballou WR, Greenwood B, Tanner M, Cohen J, Kremsner PG, Lell B, Owusu-Agyei S, Abdulla S. Evaluation of the safety and immunogenicity of the RTS,S/AS01E malaria candidate vaccine when integrated in the expanded program of immunization. J Infect Dis. 2010 Oct 1;202(7):1076-87. doi: 10.1086/656190. PMID 20735271
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 106369 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 106369 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 106369 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 106369 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 106369 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 106369 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study comprised a vaccination phase (Months 0-8) and a follow-up phase (Months 8-19). The Stamaril™ vaccine was not part of the EPI Tanzanian vaccination schedule at study planning. Hence this vaccine was not administered to subjects from Tanzania.
Period: Overall Study
Arm/Group | GSK 257049 1 Group | GSK 257049 2 Group | Tritanrix™ HepB/Hiberix™ Group
Started | 170 | 170 | 171
Completed | 151 | 156 | 148
Not Completed | 19 | 14 | 23
Not completed — Withdrawal by Subject | 5 | 3 | 4
Not completed — Lost to Follow-up | 14 | 10 | 13
Not completed — Physician Decision | 0 | 0 | 2
Not completed — Death | 0 | 1 | 3
Not completed — Other | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK 257049 1 Group | GSK 257049 2 Group | Tritanrix™ HepB/Hiberix™ Group | Total
Number analyzed (Participants) | 170 | 170 | 171 | 511
Age, Continuous [Mean (Standard Deviation); unit: Weeks] | 7.0 (0.97) | 7.1 (1.05) | 7.0 (0.97) | 7.0 (1.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90 | 84 | 78 | 252
  Male | 80 | 86 | 93 | 259
Region of Enrollment [Number; unit: Subjects]
  Gabon | 73 | 73 | 74 | 220
  Ghana | 27 | 27 | 27 | 81
  Tanzania | 70 | 70 | 70 | 210

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Serious Adverse Events (SAEs).
Description: SAEs were defined as medical occurrences that resulted in death, were life threatening, required hospitalization or prolongation of hospitalization or resulted in disability/incapacity.
Time Frame: From Month 0 to Month 8
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Number; unit: subjects
Arm/Group | GSK 257049 1 Group | GSK 257049 2 Group | Tritanrix™ HepB/Hiberix™ Group
Number analyzed (Participants) | 170 | 170 | 171
subjects | 38 | 28 | 33

2. Secondary Outcome: Concentrations of Antibodies Against Hepatitis B (Anti-HB Antibodies).
Description: Anti-HB antibody concentrations were expressed as geometric mean concentrations (GMCs) in milli-international unit per milliliter (mIU/mL). The seroprotection assay cut-off was 10 mIU/mL. This outcome only covers results for the GSK 257049 1 Group.
Time Frame: At Months 0, 1, 3 and 7.
Population: The analysis was performed on the According-to-Protocol cohort for immunogenicity, which included all evaluable subjects (i.e. those meeting all eligibility criteria, complying with the procedures defined in the protocol, with no elimination criteria during the study) for whom data concerning immunogenicity endpoint measures were available.
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | GSK 257049 1 Group
Number analyzed (Participants) | 145
mIU/mL
  Anti-HB, Month 0 [N=145] | 12.5 [9.9 to 15.7]
  Anti-HB, Month 1 [N=133] | 173.4 [131.9 to 228.0]
  Anti-HB, Month 3 [N=130] | 1355.7 [1100.6 to 1669.9]
  Anti-HB, Month 7 [N=137] | 1555.5 [1315.8 to 1839.0]

3. Secondary Outcome: Concentrations of Antibodies Against Hepatitis B (Anti-HB Antibodies).
Description: Anti-HB antibody concentrations were expressed as geometric mean concentrations (GMCs) in milli-international unit per milliliter (mIU/mL). The seroprotection assay cut-off was 10 mIU/mL. This outcome only covers results for the GSK 257049 2 Group.
Time Frame: At Months 0, 3, 7 and 8.
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | GSK 257049 2 Group
Number analyzed (Participants) | 131
mIU/mL
  Anti-HB, Month 0 [N=131] | 9.6 [7.8 to 11.8]
  Anti-HB, Month 3 [N=119] | 651.2 [541.1 to 783.8]
  Anti-HB, Month 7 [N=126] | 1133.1 [972.3 to 1320.6]
  Anti-HB, Month 8 [N=125] | 59813.5 [47050.5 to 76038.6]

4. Secondary Outcome: Concentrations of Antibodies Against Hepatitis B (Anti-HB Antibodies).
Description: Anti-HB antibody concentrations were expressed as geometric mean concentrations (GMCs) in milli-international unit per milliliter (mIU/mL). The seroprotection assay cut-off was 10 mIU/mL. This outcome only covers results for the Tritanrix™ HepB/Hiberix™ Group.
Time Frame: At Months 0, 3, 7 and 8.
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Tritanrix™ HepB/Hiberix™ Group
Number analyzed (Participants) | 143
mIU/mL
  Anti-HB, Month 0 [N=143] | 8.7 [7.3 to 10.5]
  Anti-HB, Month 3 [N=126] | 338.0 [266.3 to 429.0]
  Anti-HB, Month 7 [N=131] | 159.9 [127.0 to 201.3]
  Anti-HB, Month 8 [N=133] | 162.4 [127.9 to 206.3]

5. Secondary Outcome: Concentrations of Anti-diphtheria (Anti-D) and Anti-tetanus (Anti-T) Antibodies.
Description: Anti-D and Anti-T antibody concentrations were expressed as geometric mean concentrations (GMCs) in international unit per milliliter (IU/mL). The seroprotection assay cut-off was 0.1 IU/mL.
Time Frame: At Month 3
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | GSK 257049 1 Group | GSK 257049 2 Group | Tritanrix™ HepB/Hiberix™ Group
Number analyzed (Participants) | 142 | 133 | 142
IU/mL
  Anti-D | 1.0 [0.9 to 1.2] | 1.1 [0.9 to 1.3] | 1.4 [1.2 to 1.7]
  Anti-T | 2.8 [2.3 to 3.3] | 2.6 [2.2 to 3.1] | 3.7 [3.2 to 4.3]

6. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs).
Description: as for outcome 1
Time Frame: From Month 8 to Month 19
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Number; unit: subjects
Arm/Group | GSK 257049 1 Group | GSK 257049 2 Group | Tritanrix™ HepB/Hiberix™ Group
Number analyzed (Participants) | 170 | 170 | 171
subjects | 28 | 24 | 27

7. Secondary Outcome: Concentrations of Anti-polyribosyl Ribitol Phosphate (Anti-PRP) Antibodies.
Description: Anti-PRP antibody concentrations were expressed as geometric mean concentrations (GMCs) in microgram per milliliter (µg/mL). The seroprotection assay cut-off was 0.15 µg/mL.
Time Frame: At Month 3
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | GSK 257049 1 Group | GSK 257049 2 Group | Tritanrix™ HepB/Hiberix™ Group
Number analyzed (Participants) | 141 | 132 | 142
µg/mL | 13.3 [10.5 to 16.7] | 15.7 [12.6 to 19.4] | 18.6 [14.8 to 23.5]

8. Secondary Outcome: Titers for Antibodies Against Poliomyelitis Types 1, 2 and 3 (Anti-Polio 1, 2 and 3 Antibodies).
Description: Anti-Polio 1, 2 and 3 antibody titers were expressed as geometric mean titers (GMTs). The seroprotection assay cut-off was 8.
Time Frame: At Month 3
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | GSK 257049 1 Group | GSK 257049 2 Group | Tritanrix™ HepB/Hiberix™ Group
Number analyzed (Participants) | 136 | 125 | 133
titers
  Anti-Polio 1 [N=136;125;131] | 463.6 [342.8 to 627.0] | 485.5 [342.5 to 688.3] | 500.0 [365.0 to 684.9]
  Anti-Polio 2 [N=135;124;131] | 494.0 [389.7 to 626.2] | 563.2 [457.3 to 693.6] | 406.8 [329.1 to 502.9]
  Anti-Polio 3 [N=135;125;133] | 123.5 [92.1 to 165.6] | 148.7 [112.2 to 197.0] | 205.1 [156.5 to 268.7]

9. Secondary Outcome: Concentrations of Anti-Bordetella Pertussis Toxin (Anti-BPT) Antibodies.
Description: Anti-BPT antibodies were measured by enzyme-linked immunosorbent assay (ELISA). Concentrations were expressed as geometric mean concentrations (GMCs) in ELISA unit per milliliter (EL.U/mL). The seropositivity assay cut-off was 15 EL.U/mL.
Time Frame: At Month 3
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | GSK 257049 1 Group | GSK 257049 2 Group | Tritanrix™ HepB/Hiberix™ Group
Number analyzed (Participants) | 139 | 131 | 139
EL.U/mL | 85.3 [76.8 to 94.6] | 104.4 [94.8 to 115.0] | 106.5 [96.1 to 118.1]

10. Secondary Outcome: Concentrations of Anti-measles Antibodies.
Description: Anti-measles antibody concentrations were expressed as geometric mean concentrations (GMCs) in milli-international unit per milliliter (mIU/mL). The seropositivity assay cut-off was 150 mIU/mL. The analysis was only performed on subjects from the GSK 257049 2 and Tritanrix™ HepB/Hiberix™ groups.
Time Frame: At Months 7 and 8.
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | GSK 257049 2 Group | Tritanrix™ HepB/Hiberix™ Group
Number analyzed (Participants) | 119 | 122
mIU/mL
  Anti-measles, Month 7 [N=112;120] | 75.0 [75.0 to 75.0] | 1295.2 [1052.1 to 1594.5]
  Anti-measles, Month 8 [N=119;122] | 76.2 [73.8 to 78.6] | 1299.0 [1038.8 to 1624.4]

11. Secondary Outcome: Titers for Anti-yellow Fever Antibodies.
Description: Anti-yellow fever antibody titers were expressed as geometric mean titers (GMTs). The seroprotection assay cut-off was 10. The analysis was only performed on subjects from the GSK 257049 2 and Tritanrix™ HepB/Hiberix™ groups.
  The analysis was only performed on subjects from the GSK 257049 2 and Tritanrix™ HepB/Hiberix™ groups.
Time Frame: At Months 7 and 8.
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | GSK 257049 2 Group | Tritanrix™ HepB/Hiberix™ Group
Number analyzed (Participants) | 62 | 64
titers
  Anti-yellow fever, Month 7 [N=41;62] | 5.3 [4.8 to 5.8] | 5.9 [5.1 to 6.9]
  Anti-yellow fever, Month 8 [N=46;64] | 172.2 [135.9 to 236.3] | 183.4 [134.0 to 250.9]

12. Secondary Outcome: Concentrations of Anti-circumsporozoite Protein (Anti-CS) Antibodies.
Description: Anti-CS antibody antibodies were measured by enzyme-linked immunosorbent assay (ELISA). Concentrations were expressed as geometric mean concentrations (GMCs) in ELISA unit per milliliter (EL.U/mL). The seropositivity assay cut-off was 0.5 EL.U/mL. This outcome only covers results for the GSK 257049 1 Group.
Time Frame: At Months 0, 1, 3 and 7.
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | GSK 257049 1 Group
Number analyzed (Participants) | 153
EL.U/mL
  Anti-CS, Month 0 [N=153] | 0.4 [0.3 to 0.4]
  Anti-CS, Month 2 [N=137] | 86.6 [66.5 to 112.7]
  Anti-CS, Month 3 [N=131] | 190.3 [154.3 to 234.7]
  Anti-CS, Month 7 [N=137] | 35.3 [28.5 to 43.8]

13. Secondary Outcome: Concentrations of Anti-circumsporozoite Protein (Anti-CS) Antibodies.
Description: Anti-CS antiibodies were measured by enzyme-linked immunosorbent assay (ELISA). Concentrations were expressed as geometric mean concentrations (GMCs) in ELISA unit per milliliter (EL.U/mL). The seropositivity assay cut-off was 0.5 EL.U/mL. This outcome only covers results for the GSK 257049 2 Group.
Time Frame: At Months 0, 3, 7 and 8.
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | GSK 257049 2 Group
Number analyzed (Participants) | 141
EL.U/mL
  Anti-CS, Month 0 [N=141] | 0.4 [0.3 to 0.4]
  Anti-CS, Month 3 [N=121] | 57.7 [43.7 to 76.2]
  Anti-CS, Month 7 [N=127] | 6.1 [4.6 to 7.9]
  Anti-CS, Month 8 [N=127] | 107.8 [81.1 to 143.4]

14. Secondary Outcome: Concentrations of Anti-circumsporozoite Protein (Anti-CS) Antibodies.
Description: Anti-CS antibodies were measured by Enzyme-linked immunosorbent assay (ELISA). Concentrations were expressed as geometric mean concentrations (GMCs) in ELISA unit per milliliter (EL.U/mL). The seropositivity assay cut-off was 0.5 EL.U/mL. This outcome only covers results for the Tritanrix™ HepB/Hiberix™ Group.
Time Frame: At Months 0, 3, 7 and 8.
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Tritanrix™ HepB/Hiberix™ Group
Number analyzed (Participants) | 156
EL.U/mL
  Anti-CS, Month 0 [N=156] | 0.4 [0.3 to 0.4]
  Anti-CS, Month 3 [N=129] | 0.3 [0.3 to 0.3]
  Anti-CS, Month 7 [N=132] | 0.3 [0.3 to 0.3]
  Anti-CS, Month 8 [N=135] | 0.3 [0.3 to 0.3]

15. Secondary Outcome: Number of Subjects With Solicited Local Symptoms.
Description: Assessed solicited local symptoms were pain and swelling at injection site following vaccination with each of the following study vaccines administered intramuscularly, e. a. the Tritanrix™ HepB/Hib, Rouvax™, GSK 257049 and Stamaril™ vaccines. The numbers of subjects with each of the assessed solicited local symptoms reported were tabulated for each vaccine administered, separately.
Time Frame: During the 7-day (Days 0-6) follow-up period after any vaccination with the Tritanrix™ HepB/Hib, Rouvax™, GSK 257049 and Stamaril™ vaccines.
Population: The Total Vaccinated cohort included all vaccinated subjects whose symptom sheet was completed.
Measure: Number; unit: subjects
Arm/Group | GSK 257049 1 Group | GSK 257049 2 Group | Tritanrix™ HepB/Hiberix™ Group
Number analyzed (Participants) | 170 | 170 | 171
subjects
  Pain - GSK 257049 [N=170;170;0] | 126 | 116 | NA — The GSK 257049 vaccine was not administered to subjects from the Tritanrix™ HepB/Hiberix™ Group group.
  Swelling - GSK 257049 [N=170;170;0] | 28 | 44 | NA — The GSK 257049 vaccine was not administered to subjects from the Tritanrix™ HepB/Hiberix™ Group group.
  Pain - Rouvax™ [N=163;161;159] | 52 | 54 | 47
  Swelling - Rouvax™ [N=163;161;159] | 20 | 21 | 16
  Pain - Stamaril™ [N=95;94;94] | 2 | 7 | 2
  Swelling - Stamaril™ [N=95;94;94] | 0 | 1 | 0
  Pain - Tritanrix™ HepB/Hib [N=170;170;171] | 127 | 133 | 140
  Swelling - Tritanrix™ HepB/Hib [N=170;170;171] | 47 | 68 | 68

16. Secondary Outcome: Number of Subjects With Solicited General Symptoms.
Description: Assessed solicited general symptoms were drowsiness, fever [axillary temperature equal or above (≥) 37.5 degrees Celsius (°C)], irritability and loss of appetite following any vaccination with any of the study vaccines, e. a. the Tritanrix™ HepB/Hib, Rouvax™, GSK 257049, Stamaril™ and Polio Sabin™ vaccines.
Time Frame: During the 7-day (Days 0-6) follow-up period after any vaccination
Population: The Total Vaccinated cohort included all vaccinated subjects whose symptom sheet was completed.
Measure: Number; unit: subjects
Arm/Group | GSK 257049 1 Group | GSK 257049 2 Group | Tritanrix™ HepB/Hiberix™ Group
Number analyzed (Participants) | 170 | 170 | 171
subjects
  Drowsiness | 82 | 97 | 72
  Fever (axillary temperature ≥ 37.5°C) | 102 | 95 | 75
  Irritability | 124 | 131 | 118
  Loss of appetite | 68 | 83 | 70

17. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs)
Description: An unsolicited AE is any AE (i.e. any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with use of a medicinal product, whether or not considered related to the medicinal product) reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Unsolicited AEs were assessed following vaccination with any of the study vaccines, e. a. the Tritanrix™ HepB/Hib, Rouvax™, GSK 257049, Stamaril™ and Polio Sabin™ vaccines.
Time Frame: During the 30-day (Days 0-29) follow-up period after any vaccination
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Number; unit: subjects
Arm/Group | GSK 257049 1 Group | GSK 257049 2 Group | Tritanrix™ HepB/Hiberix™ Group
Number analyzed (Participants) | 170 | 170 | 171
subjects | 160 | 161 | 164

18. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs).
Description: as for outcome 1
Time Frame: From Month 0 to Month 19
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects.
Measure: Number; unit: subjects
Arm/Group | GSK 257049 1 Group | GSK 257049 2 Group | Tritanrix™ HepB/Hiberix™ Group
Number analyzed (Participants) | 170 | 170 | 171
subjects | 57 | 47 | 49

ADVERSE EVENTS:
Time Frame: SAEs: entire study period (Months 0-19); Solicited local/general symptoms and Unsolicited AEs: during the 7- and 30-day (Days 0-29) post-vaccination period, respectively.
Description: 3 subjects in the Tritanrix™ HepB/Hiberix™ Group died after experiencing SAEs (malnutrition (Months 0-8), and Acquired immunodeficiency syndrome, Pneumonia and Sepsis (Months 8-19)). None was assessed by the investigator to be related to study vaccines.
Arm/Group | GSK 257049 1 Group | GSK 257049 2 Group | Tritanrix™ HepB/Hiberix™ Group
Serious Adverse Events (participants affected / at risk) | 57/170 | 47/170 | 49/171
Other Adverse Events (participants affected / at risk) | 169/170 | 169/170 | 171/171
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK 257049 1 Group (N=170) | GSK 257049 2 Group (N=170) | Tritanrix™ HepB/Hiberix™ Group (N=171)
Gastroenteritis (Infections and infestations) | 17 | 10 | 14 — SAE reported between Month 0 and Month 8.
Plasmodium falciparum infection (Infections and infestations) | 5 | 10 | 13 — SAE reported between Month 0 and Month 8.
Pneumonia (Infections and infestations) | 11 | 9 | 8 — SAE reported between Month 0 and Month 8.
Anaemia (Blood and lymphatic system disorders) | 6 | 10 | 10 — SAE reported between Month 0 and Month 8.
Upper respiratory tract infection (Infections and infestations) | 5 | 4 | 4 — SAE reported between Month 0 and Month 8.
Impetigo (Infections and infestations) | 4 | 0 | 3 — SAE reported between Month 0 and Month 8.
Sepsis (Infections and infestations) | 2 | 2 | 3 — SAE reported between Month 0 and Month 8.
Febrile convulsion (Nervous system disorders) | 1 | 4 | 0 — SAE reported between Month 0 and Month 8.
Urinary tract infection (Infections and infestations) | 3 | 2 | 0 — SAE reported between Month 0 and Month 8.
Otitis media (Infections and infestations) | 3 | 0 | 1 — SAE reported between Month 0 and Month 8.
Enteritis (Gastrointestinal disorders) | 1 | 1 | 1 — SAE reported between Month 0 and Month 8.
Acarodermatitis (Infections and infestations) | 0 | 0 | 2 — SAE reported between Month 0 and Month 8.
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 — SAE reported between Month 0 and Month 8.
Bronchitis (Infections and infestations) | 1 | 1 | 0 — SAE reported between Month 0 and Month 8.
Bronchopneumonia (Infections and infestations) | 1 | 1 | 0 — SAE reported between Month 0 and Month 8.
Escherichia urinary tract infection (Infections and infestations) | 1 | 1 | 0 — SAE reported between Month 0 and Month 8.
Salmonella sepsis (Infections and infestations) | 1 | 1 | 0 — SAE reported between Month 0 and Month 8.
Sickle cell anaemia (Congenital, familial and genetic disorders) | 1 | 1 | 0 — SAE reported between Month 0 and Month 8.
Sickle cell anaemia with crisis (Congenital, familial and genetic disorders) | 1 | 1 | 0 — SAE reported between Month 0 and Month 8.
Acquired immunodeficiency syndrome (Infections and infestations) | 0 | 0 | 1 — SAE reported between Month 0 and Month 8.
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 — SAE reported between Month 0 and Month 8.
Blepharitis (Eye disorders) | 1 | 0 | 0 — SAE reported between Month 0 and Month 8.
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 — SAE reported between Month 0 and Month 8.
Cataract congenital (Congenital, familial and genetic disorders) | 0 | 0 | 1 — SAE reported between Month 0 and Month 8.
Conjunctivitis (Eye disorders) | 0 | 1 | 0 — SAE reported between Month 0 and Month 8.
Convulsion (Nervous system disorders) | 0 | 0 | 1 — SAE reported between Month 0 and Month 8.
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 — SAE reported between Month 0 and Month 8.
Extrapulmonary tuberculosis (Infections and infestations) | 0 | 1 | 0 — SAE reported between Month 0 and Month 8.
Hydrocele male infected (Infections and infestations) | 1 | 0 | 0 — SAE reported between Month 0 and Month 8.
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 1 — SAE reported between Month 0 and Month 8.
Mastoiditis (Infections and infestations) | 0 | 0 | 1 — SAE reported between Month 0 and Month 8.
Microcytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 — SAE reported between Month 0 and Month 8.
Otitis media acute (Infections and infestations) | 0 | 1 | 0 — SAE reported between Month 0 and Month 8.
Periorbital abscess (Infections and infestations) | 1 | 0 | 0 — SAE reported between Month 0 and Month 8.
Pharyngitis (Infections and infestations) | 0 | 1 | 0 — SAE reported between Month 0 and Month 8.
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 — SAE reported between Month 0 and Month 8.
Pyrexia (General disorders) | 1 | 0 | 0 — SAE reported between Month 0 and Month 8.
Rhinitis (Infections and infestations) | 0 | 1 | 0 — SAE reported between Month 0 and Month 8.
Skin infection (Infections and infestations) | 1 | 0 | 0 — SAE reported between Month 0 and Month 8.
Plasmodium falciparum infection (Infections and infestations) | 6 | 6 | 14 — SAE reported between Month 8 and Month 19.
Anaemia (Blood and lymphatic system disorders) | 6 | 6 | 10 — SAE reported between Month 8 and Month 19.
Pneumonia (Infections and infestations) | 5 | 7 | 7 — SAE reported between Month 8 and Month 19.
Upper respiratory tract infection (Infections and infestations) | 7 | 4 | 5 — SAE reported between Month 8 and Month 19.
Gastroenteritis (Infections and infestations) | 7 | 6 | 2 — SAE reported between Month 8 and Month 19.
Impetigo (Infections and infestations) | 1 | 3 | 3 — SAE reported between Month 8 and Month 19.
Bronchitis (Infections and infestations) | 3 | 2 | 1 — SAE reported between Month 8 and Month 19.
Malnutrition (Metabolism and nutrition disorders) | 2 | 1 | 1 — SAE reported between Month 8 and Month 19.
Urinary tract infection (Infections and infestations) | 3 | 0 | 1 — SAE reported between Month 8 and Month 19.
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 — SAE reported between Month 8 and Month 19.
Sepsis (Infections and infestations) | 1 | 0 | 2 — SAE reported between Month 8 and Month 19.
Bronchopneumonia (Infections and infestations) | 1 | 1 | 0 — SAE reported between Month 8 and Month 19.
Convulsion (Nervous system disorders) | 1 | 0 | 1 — SAE reported between Month 8 and Month 19.
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1 — SAE reported between Month 8 and Month 19.
Febrile convulsion (Nervous system disorders) | 0 | 2 | 0 — SAE reported between Month 8 and Month 19.
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 — SAE reported between Month 8 and Month 19.
Nasopharyngitis (Infections and infestations) | 0 | 0 | 2 — SAE reported between Month 8 and Month 19.
Otitis media (Infections and infestations) | 1 | 0 | 1 — SAE reported between Month 8 and Month 19.
Sickle cell anaemia with crisis (Congenital, familial and genetic disorders) | 1 | 1 | 0 — SAE reported between Month 8 and Month 19.
Thermal burn (Injury, poisoning and procedural complications) | 2 | 0 | 0 — SAE reported between Month 8 and Month 19.
Accidental exposure (Injury, poisoning and procedural complications) | 1 | 0 | 0 — SAE reported between Month 8 and Month 19.
Acquired immunodeficiency syndrome (Infections and infestations) | 0 | 0 | 1 — SAE reported between Month 8 and Month 19.
Dysentery (Infections and infestations) | 1 | 0 | 0 — SAE reported between Month 8 and Month 19.
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 1 — SAE reported between Month 8 and Month 19.
Glomerulonephritis (Renal and urinary disorders) | 0 | 0 | 1 — SAE reported between Month 8 and Month 19.
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 — SAE reported between Month 8 and Month 19.
Otitis media acute (Infections and infestations) | 0 | 0 | 1 — SAE reported between Month 8 and Month 19.
Otitis media chronic (Infections and infestations) | 0 | 1 | 0 — SAE reported between Month 8 and Month 19.
Petroleum distillate poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 1 — SAE reported between Month 8 and Month 19.
Pharyngitis (Infections and infestations) | 0 | 1 | 0 — SAE reported between Month 8 and Month 19.
Pneumonitis chemical (Injury, poisoning and procedural complications) | 0 | 1 | 0 — SAE reported between Month 8 and Month 19.
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 — SAE reported between Month 8 and Month 19.
Pyrexia (General disorders) | 1 | 0 | 0 — SAE reported between Month 8 and Month 19.
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 — SAE reported between Month 8 and Month 19.
Skin infection (Infections and infestations) | 0 | 0 | 1 — SAE reported between Month 8 and Month 19.
Urinary tract infection pseudomonal (Infections and infestations) | 0 | 1 | 0 — SAE reported between Month 8 and Month 19.
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 — SAE reported between Month 8 and Month 19.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | GSK 257049 1 Group (N=170) | GSK 257049 2 Group (N=170) | Tritanrix™ HepB/Hiberix™ Group (N=171)
Drowsiness (General disorders) | 82 | 97 | 72
Fever (General disorders) | 102 | 95 | 75
Irritability (General disorders) | 124 | 131 | 118
Loss of appetite (General disorders) | 68 | 83 | 70
Pain (General disorders) | 127 | 133 | 140 — Solicited local symptom reported after vaccination with Tritanrix™ HepB/Hib
Pain (General disorders) | 52/163 | 54/161 | 47/159 — Solicited local symptom reported after vaccination with Rouvax™.
Pain (General disorders) | 126 | 116 | 0/0 — Solicited local symptom reported after vaccination with the GSK 257049 vaccine.
Pain (General disorders) | 2/95 | 7/94 | 2/94 — Solicited local symptom reported after vaccination with Stamaril™.
Swelling (General disorders) | 47 | 68 | 68 — Solicited local symptom reported after vaccination with Tritanrix™ HepB/Hib
Swelling (General disorders) | 20/163 | 21/161 | 16/159 — Solicited local symptom reported after vaccination with Rouvax™.
Swelling (General disorders) | 28 | 44 | 0/0 — Solicited local symptom reported after vaccination with the GSK 257049 vaccine
Upper respiratory tract infection (Infections and infestations) | 66 | 66 | 65
Nasopharyngitis (Infections and infestations) | 53 | 62 | 71
Gastroenteritis (Infections and infestations) | 29 | 25 | 32
Rhinitis (Infections and infestations) | 16 | 21 | 21
Cough (Respiratory, thoracic and mediastinal disorders) | 21 | 30 | 24
Induration (General disorders) | 26 | 28 | 29
Diarrhoea (Gastrointestinal disorders) | 21 | 24 | 24
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 19 | 19 | 23
Pneumonia (Infections and infestations) | 19 | 11 | 9
Conjunctivitis (Eye disorders) | 16 | 21 | 19
Bronchitis (Infections and infestations) | 17 | 17 | 21
Anaemia (Blood and lymphatic system disorders) | 11 | 19 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.